CLINICAL TRIAL: NCT02184260
Title: A Randomized, Multicentre, Double-blind Clinical Trial of Metamizole 2 g /8 h, I.V. Ampoules, Versus Placebo Each 8 h, I.V. Ampoules, Administered During 3 Days Consecutively as Antithermic Therapy in the Acute Phase of Ischemic Stroke. A 30-day Study. (ATIS Study)
Brief Title: Efficacy and Safety of Metamizole Versus Placebo as Antithermic Therapy in the Acute Phase of Ischemic Stroke
Acronym: ATIS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1093.15
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Dipyrone

ARMS (2):
- Metamizole (Experimental)
  Interventions: Drug: Metamizole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metamizole
  Arms: Metamizole
Drug: Placebo
  Arms: Placebo

SUMMARY:
Clinical efficacy and safety of Metamizole 2 g i.v. versus placebo, as antithermic therapy in the acute phase of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Hemispherical cerebral infarction with moderate (SSS = 30-44 points) or severe (SSS < 30 points) deficit at the time of inclusion. However, only patients with a score between 15 and 44 points on the SSS scale will be included
* Tympanic temperature between 37 and 38 degrees Celsius. The relationship between tympanic and body temperature is as follows: tympanic temperature = body temperature + 0.3 degrees Celsius
* Onset of cerebral infarction symptoms within the last 24 hours. When the time of onset of symptoms is unknown (e.g. ictus occurred while sleeping) the last time when the patient was asymptomatic will be considered as time of onset
* Normal cerebral CT scan or with signs of cerebral infarction
* Patient's written or orally witnessed informed consent in accordance with local legislation, guidelines of Good Clinical Practice (GCP) and International Conference on Harmonization (ICH)-GCP

Exclusion Criteria:

* Patients with a history of granulocytopenia, thrombocytopenia or aplastic blood diseases of any etiology. Known hypersensitivity to salicylates, pyrazolones and other nonsteroidal antiinflammatory drugs (NSAIDs). NSAID-induced bronchial asthma
* Patients with a history indicating a life expectancy less than 30 days or patients whom the investigator thinks that it will not be possible to follow for entire 30 days
* Non-cooperative
* Patients with neurological sequelae of a previous stroke
* Cerebral hemorrhage
* Pregnancy, lactation
* Participation in another clinical trial
* Intake of acetylsalicylic acid (ASA) > 300 mg per day, paracetamol or NSAIDs during the 24 hours prior to administration of the study medication
* Seizures at the start of the stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1998-12; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the functional outcome according to the Scandinavian Stroke Scale (SSS) | after 30 days

SECONDARY OUTCOMES:
Assessment of functional outcome according to SSS | Baseline, after 3 and 7 days
Number of patients with score of SSS < 30 points | after 30 days
Clinical impression assessed on the Modified Rankin Scale | after 30 days
Effect on the activities of daily living assessed on Barthel Index | after 30 days
Number of patients requiring rescue therapy | up to 30 days
Duration of hospital stay | up to 30 days
Assessment of tympanic temperature | up to 3 days after start of treatment
Percentage of mortality | after 30 days
Number of patients with adverse events | up to 30 days